CLINICAL TRIAL: NCT04122183
Title: Internet Auditory Rehabilitation: Innovative Follow-up to Adult Hearing Screening.
Brief Title: Internet Auditory Rehabilitation: Follow-up to Adult Hearing Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: William Demant Foundation (Formerly known as the Oticon Foundation) (Unknown)
Responsible Party: Principal Investigator, Laura N. Galloway, Lecturer, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.0663
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Hearing Loss
Keywords: Hearing Screening, Auditory Rehabilitation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program Group (Experimental): Following a failed hearing screening, participants will be offered the standard of care (information sheet recommending a comprehensive hearing evaluation) and asked to complete the iManage Program. Six months after the screening participants will be asked if they visited an audiologist.
  Interventions: Other: iManage (my hearing loss)
- Delayed Program Group (No Intervention): Following a failed hearing screening, participants will be offered the standard of care (information sheet recommending a comprehensive hearing evaluation). Six months after the screening participants will be asked if they visited an audiologist and they will be given the opportunity to complete the iManage Program.

INTERVENTIONS:
Other: iManage (my hearing loss) — An internet-based decision coaching guide to help an individual decide if they wish to visit an audiologist.
  Arms: Program Group

SUMMARY:
The purpose of this study is to see if a newly developed program called "I Manage my hearing loss" (iManage) will increase the number of individuals who visit an audiologist after failing a hearing screening. The iManage program will educate individuals about hearing loss, demonstrate that hearing problems are important, demonstrate that support from family and friends is important and help participants identify the benefits and concerns related to seeking help for hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Subject must fail a hearing screening (any threshold >34 decibels hearing level at 2000 or 3000 Hertz in either ear) or show equivalent or greater degree of hearing loss on most recent audiogram.
* Free of obvious outer or middle ear disease (as measured by otoscopy)
* Between the ages of 45 and 85
* Pass a health literacy screening
* Pass a thinking skills screening

Exclusion Criteria:

* Experience seeing an audiologist for a hearing evaluation or management
* Experience using a hearing aid

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Audiologist visit | 6 months following the failed hearing screening
  The percentage of individuals who visit an audiologist for a comprehensive hearing evaluation.

SECONDARY OUTCOMES:
Change on the Health Belief Questionnaire, a survey that measures attitudes about the 6 constructs of the Health Belief Model as related to seeking hearing healthcare | Baseline (within one week of screening) and 6 months post baseline
  Mean score (which can range between 1 and 11) on each of 6 scales: perceived susceptibility, perceived severity, perceived benefits, perceived barriers, perceived self-efficacy, and cues to action. A higher score indicates greater agreement with the construct.
Change on the Readiness for Change Questionnaire, a single-item questionnaire that attempts to place the participant on a continuum regarding readiness for hearing healthcare as outline by the Transtheoretical Model. | Baseline, 4 weeks post baseline, and 6 months post baseline
  Participants will select the statement that best describes their view of their hearing status, 1 indicates "precontemplation", 2 indicates "contemplation", 3 indicates, "preparation", 4 indicates "action" on the Transtheoretical Model Continuum.
Total score on the Hearing Loss Support Scale, a questionnaire that measures self-perceived informational and emotional support from family, peers, and healthcare providers about managing hearing loss. | Baseline, and 6 months post baseline
  Total score can range between 7 and 49, with a higher score indicating greater support from others.

OTHER OUTCOMES:
Program uptake | 3 months following the failed hearing screening
  Percentage of experimental participants who begin the iManage program
Program completion | 3 months following the failed hearing screening
  Percentage of experimental participants who complete the iManage program
Mean scores on the Audiology Decision Making Scale, a scale designed to measure preparedness for decision making for 13 specific decision processes | 4 weeks after completion of iManage Program
  Mean score can range between 1 and 5 with higher scores indicating greater self-perceived usefulness of the iManage Program in making a decision about hearing healthcare.
A focus group of individuals who completed the iManage program to learn participants perceptions about the content, benefits and drawbacks of the iManage program | 6 to 8 weeks after completion of iManage Program
  Qualitative thematic analysis will indicate common attitudes (themes) about the iManage program

CONTACTS AND LOCATIONS:
Overall Officials: Laura Galloway, AuD, Principal Investigator — Professor
Locations (1):
- University of Louisville, Program in Audiology, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is no individual participant data (IPD) sharing plan at this time as this is a feasibility study.